CLINICAL TRIAL: NCT05124600
Title: An Individualized-health eLibrary App for People With Multiple Sclerosis: Testing Feasibility and Effectiveness of a Brief Education Intervention
Brief Title: An Individualized-health eLibrary App for People With Multiple Sclerosis
Acronym: SavvyHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Chung-Yi Chiu, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20117; RB19148 (Other Grant/Funding Number: University of Illinois Urbana-Champaign)
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: eHealth; mHealth
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SavvyHealth (Experimental): Participants will use the new app, SavvyHealth, for 21 days.
  Interventions: Device: SavvyHealth
- Waiting list (No Intervention): Participants will be on the waiting list.

INTERVENTIONS:
Device: SavvyHealth — Participants will use the new app, SavvyHealth, for 21 days.
  Arms: SavvyHealth

SUMMARY:
The purpose of this study is to assess the effectiveness after using a new individualized-health e-library app named SavvyHealth among people with multiple sclerosis.

DETAILED DESCRIPTION:
Participants will use our developed app for 21 days and take a before-use survey and a post-use survey.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with MS;
* 18 years or older;
* one comorbidity evaluated by a validated comorbidity questionnaire for people with MS;
* willing to take a survey;
* willing to use the app for 21 days;
* willing to be assigned to either the intervention or control group.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MS Self-management Scale | Through study completion, an average of 1 week
  A self-reported 5-point scale, five factors: healthcare provider relationship and communication, treatment adherence, social support, MS knowledge, and health maintenance behavior.
  "Change" is being assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chungyi Chiu, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Study result report
Supporting Information: CSR